CLINICAL TRIAL: NCT00133510
Title: Prospective Comparative Study of the Humoral and Cell-Mediated Immune Responses to the Trivalent Subviron Influenza Vaccine in Pediatric Liver Transplant Recipients as an Indicator for Response of Immunocompromised Subjects to Vaccination Against Agents of Bioterrorism
Brief Title: Influenza Vaccine in Pediatric Transplant Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 04-050
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2008-03

CONDITIONS: Influenza
Keywords: children, immunocompromised, influenza, liver transplant
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Trivalent Subviron Influenza vaccine (Fluzone)

SUMMARY:
The purpose of this study is to evaluate how well children responds to the recommended trivalent subviron influenza vaccine (flu shot). Children who have had a liver transplant and receive their post-transplant care at Mount Sinai and their siblings are being invited to participate in this study. Study procedures will include a review of medical records, physical examination, and up to 2 flu shots. All participants will receive the flu vaccine. Four weeks after the first flu shot, participants will return to the clinic for a physical exam, blood sample collection, and a second flu shot as recommended. Following each vaccination, parents will be asked to record their children's temperatures and any experienced side effects in a diary card for two weeks. Participants will be involved in study related procedures for up to 8 months.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the humoral and cell-mediated immune response to the trivalent subviron influenza vaccine in pediatric liver transplant recipients. Additionally, researchers will attempt to correlate the humoral and cell-mediated immune response with parameters that may predict a subject's ability to respond to the vaccine, such as time from transplant, immunosuppressive agents, previous episodes of rejection or cytomegalovirus infection, T-cell numbers and T-cell responses to mitogens or antigens. Understanding the immune response to influenza will provide insight not only into the response to the trivalent subviron influenza vaccine but to other vaccines being developed against agents of bioterrorism, in particular those that may use influenza or related viruses as a backbone. This is a single center, prospective comparative study of the humoral and cell-mediated immune responses to the trivalent subviron influenza vaccine for the 2004-2005 and 2005-2006 influenza seasons in outpatient pediatric liver transplant recipients and their healthy siblings. There are two study arms, the liver transplant recipients (n=44) and the healthy controls (n=22). All study subjects will receive the vaccine at enrollment. Enrollment into this study will be extended into the 2005-2006 influenza season. The trivalent subviron influenza vaccine for the 2005-2006 influenza season will differ from that for the 2004-2005 influenza season with respect to the H3N2 viral strains. The cell-mediated and humoral immune responses of patients to the two H3N2 viral strains will be analyzed together and separately to assess potential differences in immunogenicity between the two viral strains. Humoral and cell-mediated immune responses will be obtained at baseline and following immunization. Healthy siblings are used as controls to ensure equal burden of influenza disease among study participants. Participants will be involved in study related procedures for up to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parent/guardian and assent from participants, when applicable, must have been obtained and signed freely.
* Between the ages of 6 months and 17 years.
* Three months have elapsed since liver transplantation.
* Recipient of a liver transplant or live with a sibling who is the recipient of a liver transplant.
* Must have the ability to comply with the study procedures for the entire length of the study.

Exclusion Criteria:

* Previous immunization with an influenza vaccine for the 2004-2005 or 2005-2006 influenza season.
* Known hypersensitivity reaction to the vaccine or vaccine component including eggs or gelatin.
* History of Guillian-Barré syndrome.
* Receipt of an immunoglobulin product (including intravenous or intramuscular immunoglobulin preparations, cytomegalovirus hyperimmunoglobulin and varicella-zoster immunoglobulin) within 3 months of vaccination.
* Receipt of any live viral vaccines within 4 weeks or an inactivated viral vaccine within 2 weeks of enrollment.
* Subjects who have experienced an acute febrile illness within the preceding 48 hours will have immunization deferred and be rescheduled once their fever has resolved.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2004-11; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, New York, New York, United States